CLINICAL TRIAL: NCT04240678
Title: The Effect of an Electronic Medical Record (EMR) Alert on Hepatitis B Screening: A Randomized Controlled Trial
Brief Title: The Effect of an Electronic Medical Record (EMR) Alert on Hepatitis B Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 8301387
Record Dates: First submitted 2020-01-17; First posted 2020-01-27 (Actual); Results first posted 2021-02-26 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis B
Keywords: Mass Screening
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBV Alert Group (Experimental)
  Interventions: Other: Electronic HBV Alert
- Control Group (No Intervention)

INTERVENTIONS:
Other: Electronic HBV Alert — Electronic HBV Alert deployed in electronic medical charts of at risk patients
  Arms: HBV Alert Group

SUMMARY:
Asian and Pacific Islander Americans at risk, but never tested for chronic hepatitis B have been randomized to receive an electronic alert in their electronic medical chart to remind primary care physicians to screen them for chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria: Asian and Pacific Islanders (API) who have not yet received HBsAg testing. API will be identified using a novel algorithm which identifies them using their surname, language preference, country of origin.

-

Exclusion Criteria: Previous HBsAg completion.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8299 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2021-07-01 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chak E, Li CS, Chen MS Jr, MacDonald S, Bowlus C. Electronic health record alerts enhance mass screening for chronic hepatitis B. Sci Rep. 2020 Nov 5;10(1):19153. doi: 10.1038/s41598-020-75842-8. PMID 33154429

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: No alert
Period: Overall Study
Arm/Group | HBV Alert Group | Control Group
Started | 4141 | 4158
Completed | 4141 | 4158
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients at risk for Hepatitis B
Groups:
- Total: Total of all reporting groups
Arm/Group | HBV Alert Group | Control Group | Total
Number analyzed (Participants) | 4,141 | 4,158 | 8299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4141 | 4158 | 8299
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.64 (20.88) | 51.32 (20.66) | 51.45 (20.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2,172 | 2,256 | 4428
  Male | 1,969 | 1,902 | 3871
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4,141 | 4,158 | 8299
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4,141 | 4,158 | 8299
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4,141 | 4,158 | 8299

OUTCOME MEASURES:

1. Primary Outcome: Serum Hepatitis B Surface Antigen Completion
Description: Number of patients who have completed the HBsAg test
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Alert Group | Control Group
Number analyzed (Participants) | 4,141 | 4,158
Participants | 389 | 177

2. Secondary Outcome: Serum Hepatitis B Surface Antigen Positivity
Description: Number of patients with testing positive for HBsAg
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Alert Group | Control Group
Number analyzed (Participants) | 4,141 | 4,158
Participants | 15 | 13

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | HBV Alert Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/4141 | 0/4158
Serious Adverse Events (participants affected / at risk) | 0/4141 | 0/4158
Other Adverse Events (participants affected / at risk) | 0/4141 | 0/4158

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT04240678/Prot_SAP_000.pdf